CLINICAL TRIAL: NCT02378558
Title: Phase 1 Study of Magnetic Breast Marking Clip System MagneMark
Brief Title: A Trial of a New Magnetic Breast Marking Clip
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Collaborators: MagneMark LLC (Unknown)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-03-08; MagneMark_02 (Other: maimonides)
Record Dates: First submitted 2015-02-19; First posted 2015-03-04 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Breast Neoplasms
Keywords: Breast Surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational Device (Experimental): All patients will undergo breast localization and excision of a lesion using the MagneMark system. The radiologist will insert the MagneMarker clip into the area of concern using the MagneJector device. The surgeon will then locate the MagneMaker clip using the MagneProbe. The clip and breast tissue of concern will then be removed.
  Interventions: Device: MagneMarker

INTERVENTIONS:
Device: MagneMarker — The MagneMarker system includes a magnetic clip the MagneMarker, a clip placement device the MagneJector, and a magnetic field detecting probe the MagneProbe. The MagneMarker and MagneJector are used by a radiologist during a breast localization procedure. The MagneProbe is used by a surgeon to locate the MagneMarker during breast excision.

SUMMARY:
This small pilot will allow surgeons to perform wireless breast lumpectomies using a new magnetic technology. This is a continuation of a previous project testing the technology, and the breast surgeons comfort level using this new technology.

The aim of this project is to develop a new technique for surgical excision of lesions either through surgical biopsy or lumpectomy. The current standard of care involves placing a needle then slender wire through the lesion under image guidance by a radiologist. The surgeon then removes the lesion using the wire as a guide. This new technique would place a magnet through the lesion under image guidance by a radiologist. The surgeon would then use the MagneProbe in the operating room to locate the magnet and remove the lesion. This new technique would eliminate the use of a wire that protrudes from a patient's breast. This wire is usually placed on the day of surgery, prior to the procedure. The goal of this new technique is to eliminate wire placement and increase patient comfort throughout the day of her surgery.

DETAILED DESCRIPTION:
Pilot II: Before embarking on pivotal efficacy studies, we propose a pilot II study to address the ease of transition from use of the MagneWire to fully implanted MagneMarkers. Before embarking on a pivotal study, comparing the wireless MagneMarker with a standard breast localization wire, we propose an open label single arm pilot II study. In the pilot II study each surgeon (n=3) will treat 14 cases with the MagneMarker using magnetic localization alone. The outcomes of this study will be:

1. Completeness of excision.
2. Time for the biopsy.

Overview: The goal of the MagneMark system is to replace the use of wires with the use of fully implanted MagneMarkers. In the Pilot II trial patients will be localized on the morning of their surgery comparable to the timeline utilized in a traditional wire localization procedure.

Eligibility for surgeons: Experienced breast surgeons practicing at Maimonides Medical Center with full proficiency at standard wire localized excisions as well as sentinel lymph node biopsy who have completed the required number of MagneWire guided excisions for training on the MagneMark system. Because this is a single arm pilot there will be no blinding of the surgeons involved.

Eligibility for patients: Eligible patients have a single non-palpable breast cancer (invasive or DCIS) requiring preoperative needle localization with a single wire. Lesions may include discrete solitary mammographically or sonographically identified targets that can be definitively identified by specimen imaging, including previously biopsied lesions that have been marked by a biopsy site marker. All patients who are eligible will be consented for off label use of the MagneMarker system there will be no randomization, blinding or stratification of patients.

Study Location: All procedures will be completed at the Maimonides Medical Center. Localizations will happen in the radiology suite at the Maimonides Breast Center and excisions will happen at the Ambulatory Surgery Center at Maimonides Medical Center.

Duration: For the enrolled patients participation in the trial is limited to the amount of time the localization and excision procedures take, approximately 5 hours. To enroll enough patients for three surgeons to complete fourteen surgeries we anticipate that recruitment will continue for one calendar year.

Description of device: The MagneJector will be used to insert a 1x20mm Arnokrome MagneMarker and anchor it in position with its center anchors centered in the target. Sonographic guided localizations will be performed with the MagneJector hand held while mammographic guided localizations will be performed on dedicated prone stereo tables with the MagneJector mounted on a rail. The Arnokrome component of the MagneMarker will be coated with Parylene, a plastic polymer meeting the International Organization for Standardization 10993 standards for biocompatibility.

Administration: moving through a MagneMark study procedure day.

1. On the day of the localization procedure, the patient will go to one of the three radiologist involved in the project.
2. The radiologist will insert the study device using the MagneJector.
3. The patient will be transported t the surgical suite for excision.
4. Surgery will be performed at the ambulatory surgery suite of Maimonides Medical Center.
5. The surgeon will use the MagneProbe to identify the location of the MagneMarker as well as the lesion, and remove both the MagneMarker and lesion.

Data endpoints: the rate of successful excision of the target lesion, the size and weight of the specimens removed and the presence or absence of positive tumor margins will serve as primary endpoints. Secondary endpoints will include the length of stay for the day of surgery with the hypothesis that length of stay will be significantly reduced. Additional endpoints will include comparison of the accuracy and precision of centering the marker in the center of the lesion.

ELIGIBILITY:
Inclusion Criteria:

i) Female ii) Ages 19-100 iii) Have a single breast lesion that has been previously biopsied and iv) Is discretely identified by:

1. A metallic biopsy site marker or
2. Ultrasound or
3. Mammography and v) Is scheduled for preoperative needle localization with a single wire and vi) Is English speaking vii) Is capable of making medical decisions, not cognitively impaired viii) Is being localized by a study radiologist or can be rescheduled to be localized by a study radiologist

Exclusion Criteria:

i) Cognitively impaired adults ii) Non- English speakers ii) Men

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-03; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Completeness of Excision | 1 year
  Investigators anticipate that cases using this localization and excision technique will be successful at minimum 96% of the time. The rate at which excision is successful using traditional methods. This outcome will be assessed and presented at the completion of the trial at the end of one year

SECONDARY OUTCOMES:
Time for excision | 1 year
  Investigators anticipate that cases will not take longer than traditional wire excisions. This outcome will be assessed and presented at the completion of the trial at the end of one year

CONTACTS AND LOCATIONS:
Overall Officials: Donna Marie Manasseh, MD, Principal Investigator — Chief, Division of Breast Surgery Director, Maimonides Breast Cancer Program Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided